CLINICAL TRIAL: NCT06937554
Title: Evaluation of Physical-cognitive-functional and Nutritional Parameters in Inpatients Affected by Acute Leukemia During Intensive Chemotherapy Treatment
Brief Title: Evaluation of Functional and Nutritional Parameters in Fit Acute Leukemia Patients
Acronym: FisNutEma
Status: Recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Nicola Manocchio, PhD Student, Medical Doctor, PRM Specialist, University of Rome Tor Vergata
Other Study IDs: FisNutEma
Record Dates: First submitted 2025-04-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Leukemia
Keywords: Acute leukemia; Rehabiltation; Quality of life; Nutrition
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients above 18 years, affected by Acute Leukemia, performing intensive chemotherapy
  Interventions: Other: observational follow up aimed at evaluating functional, physical, cognitive, and nutritional parameters

INTERVENTIONS:
Other: observational follow up aimed at evaluating functional, physical, cognitive, and nutritional parameters — observational follow up aimed at evaluating functional, physical, cognitive, and nutritional parameters

SUMMARY:
This single-center observational prospective longitudinal study will assess cognitive, physical, and nutritional performance in acute leukemia patients undergoing intensive chemotherapy. Patients will provide informed consent prior to enrollment. Hematologists will oversee clinical management and approve evaluations, while physical and rehabilitation medicine specialists and a nutritionist will conduct assessments. Performance will be evaluated at admission, discharge, and three weeks (21 days) after starting chemotherapy.

DETAILED DESCRIPTION:
This is an observational prospective longitudinal single-center study. All patients will be required to agree to participate in the study and to sign an informed consent prior to enrollment.

During the course of the study, the hematologists will manage the patients as per clinical practice and give clearance to perform each evaluation. All functional assessments and tests will be carried out by trained healthcare personnel with experience in the field of rehabilitation (either a Physical and Rehabilitation Medicine Resident, a Specialist, or a physiotherapist). A nutritionist will take care of assessing the nutritional aspects.

The aim of this study is to analyze the cognitive, physical and nutritional performance of AL patients hospitalized to receive intensive chemiotherapy (IC). Each item will be assessed at admission and discharge from the ward and after three weeks from the start of chemotherapy. Modifications of the considered items will be annotated and compared throughout the courses of chemotherapy, as well as relationship with indices of response and survival (Disease Free Survival, Overall Survival) will be explored. Such an effort will help further understanding how hematologic inpatients perform during IC treatment and what are the consequences on their quality of life and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patients affected by Acute Leukemia
* Inpatients performing intensive chemotherapy
* Patients with no restrictions on mobilization
* Signed written informed consent in accordance with ICH/EU/GCP guidelines and national and local laws.

Exclusion Criteria:

* Age <18 years
* Any medical condition that the attending doctor judges as limiting to perform study related tasks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Leukemia inpatients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Grip Force Test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  A grip force test using a dynamometer, also known as a handgrip dynamometer, measures how much force a person can apply with their fingers and forearms. It's a tool used to assess hand grip strength.
Modified Borg Scale (MBS) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The MBS is a subjective rating scale used to measure the intensity of physical activity. It ranges from 6 to 20 points, with 6 representing "no exertion" and 20 representing "maximal exertion." The scale is divided into four categories: 6-9 (very light), 10-12 (light), 13-15 (somewhat hard), and 16-20 (very hard). The MBS is commonly used to assess the intensity of exercise and to monitor individual responses to physical activity. It can be used by people of all ages and fitness levels
Tampa Scale of Kinesofobia (TSK) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Timed Up and Go (TUG) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  Measure of function which correlates to balance and fall risk. Start timing on the word "GO" and stop timing when the subject is seated again correctly in the chair with their back resting on the back of the chair.
  ≤ 10 seconds
  = normal
  ≤ 20 seconds
  = good mobility, can go out alone, mobile without gait aid
  ≤ 30 seconds
  = problems, cannot go outside alone, requires gait aid
  * A score of
  ≥ 14 seconds has been shown to indicate high risk of falls
Visual Analogue Scale (VAS) for pain | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).
Fatigue Severity Scale (FSS) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. A total score of less than 36 suggests that the patient may not be suffering from fatigue.
  A total score of 36 or more suggests that the patient may need further evaluation by a physician.
Functional Ambulation Classification (FAC) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. A score of 0 indicates that the patient is a non-functional ambulator (cannot walk).
  A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3).
  A score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score).
SF-12 Questionnaire | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 uses eight domains:
  Limitations in physical activities because of health problems. Limitations in social activities because of physical or emotional problems Limitations in usual role activities because of physical health problems Bodily pain General mental health (psychological distress and well-being) Limitations in usual role activities because of emotional problems Vitality (energy and fatigue) General health perceptions
Symbol Digit Modalities Test (SDMT) for processing speed | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The Symbol Digit Modalities Test (SDMT) is widely used for cognitive evaluation of information processing speed, required in many cognitive operations. The person taking the test is provided with a set of symbols, each corresponding to a number. He or she is required to write down the symbols corresponding to a series of numbers within a short space of time. The SDMT is quick (~5 min) and straightforward to administer, provides a clear test score that is not influenced by subjective interpretations on the part of the healthcare professional who administers the test, and is little affected by patients׳ age, gender or educational status.
Modified Barthel Index | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  The Modified Barthel Index is an ordinal scale which measures a person's ability to complete activities of daily living.
  The evaluated domains are:
  * Feeding
  * Bathing
  * Grooming
  * Dressing
  * Bowel
  * Bladder
  * Toilet use
  * Transfers bed-to-chair-and-back
  * Mobility on level surfaces
  * Stair negotiation The higher the score, the more independent the patient is in completing the measured activity. Higher scores also indicate the patient is more likely to return home, with varying degrees of assistance, following hospital discharge.
  The lower the score, the more dependent the patient is with the activity completion, and the more skilled care will be required at discharge.
Serum pre-albumine | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days
  Serum prealbumin levels are measured using a blood test that can help assess nutritional status. Prealbumin is a protein made in the liver that helps transport thyroid hormones and vitamin A, and controls how the body uses energy. A prealbumin level below 30 mg/dL may indicate malnutrition.
Serum albumine | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days
  A serum albumin test measures the amount of albumin in blood. Albumine dosage helps determining the presence of liver disease, kidney disease, or protein malabsorption. The normal range is 3.4 to 5.4 g/dL (34 to 54 g/L)
Body mass index (BMI) | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days
  Body mass index (BMI) is a calculation that compares a person's weight to their height. It's a screening tool that can help determine if someone is a healthy weight for their height. BMI is calculated by dividing weight in kilograms by height in meters squared.
  BMI categories:
  Underweight: BMI is below 18.5 Healthy weight: BMI is between 18.5 and 24.9 Overweight: BMI is between 25 and 29.9 Obese: BMI is between 30 and 39.9 Severely obese: BMI is 40 or higher

SECONDARY OUTCOMES:
Coin test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  For this test, subjects sit at a table and are timed as they pick up four coins (2€, 50cents, 10cents, 5cents ) and place them in a cup. They are required to pick up each coin individually.
Sock test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  Subjects sit in a standard chair. They are timed as putting on one sock
Back Scratch Test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  distance between the two middle fingers, one arm from above and one from below behind the back
Forward Bending Test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  distance between middle fingers and ground
Stability test | Initial evaluation (TO) at admission (+2 days) Intermediate evaluation (T1) at day 21 (+/- 1 day) after IC start Final evaluation (T2) at discharge (-2 days)
  subjects must stand on a single leg with eyes closed for the longest time possible while timed (max 30 seconds per limb).

CONTACTS AND LOCATIONS:
Locations (1):
- Tor Vergata university Hospital, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No